CLINICAL TRIAL: NCT04090021
Title: Genotypic Resistance-guided Triple Therapy Versus Empirical Concomitant Therapy for First-line H. Pylori Eradication.
Brief Title: Genotypic Resistance-guided Versus Empirical Therapy for H. Pylori Eradication.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Konstantopoulio-Patission General Hospital of Nea Ionia (Other)
Responsible Party: Principal Investigator, Vasilios Papastergiou, Consultant Gastroenterologist, Konstantopoulio-Patission General Hospital of Nea Ionia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10548
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Helicobacter Pylori Infection
Keywords: H. pylori; genotypic resistance; tailored therapy; concomitant therapy
MeSH Terms: interventions — Esomeprazole; Clarithromycin; Metronidazole; Amoxicillin; Levofloxacin; Rifabutin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Genotypic resistance-guided triple therapy (Experimental): In the group of genotypic resistance-guided triple therapy, a molecular assay based on DNA-strip technology was used to determine the genotypic resistance of H. Pylori to clarithromycin (23SrRNA mutations) and fluoroquinolones (gyrA mutations) from gastric biopsy specimens. According to 23SrRNA and gyrA mutational analyses, a 7-day tailored triple therapy therapy was given as follows:
  Wild-type 23SrRNA: Clarithromycin-based triple therapy comprising esomeprazole 40 mg b.i.d., amoxicillin 1 g b.i.d. and clarithromycin 500 mg b.i.d.
  23SrRNA mutated/wild-type gyrA: Levofloxacin-based triple therapy comprising esomeprazole 40 mg b.i.d., amoxicillin 1 g b.i.d. and levofloxacin 500 mg b.i.d.
  23SrRNA mutated/gyrA mutated: Rifabutin-based triple therapy comprising esomeprazole 40 mg b.i.d., amoxicillin 1 g t.i.d. and rifabutin 150 mg b.i.d.
  Interventions: Drug: Esomeprazole 40mg; Drug: Clarithromycin 500mg; Drug: Amoxicillin 1000 MG; Drug: Levofloxacin 500mg; Drug: Rifabutin 150 MG
- Empirical concomitant therapy (Active Comparator): In the empirical concomitant group, patients received esomeprazole 40mg, amoxicillin 1gr, clarithromycin 500mg and metronidazole 500mg, all b.i.d., for 10-14 days.
  Interventions: Drug: Esomeprazole 40mg; Drug: Clarithromycin 500mg; Drug: Metronidazole 500 mg; Drug: Amoxicillin 1000 MG

INTERVENTIONS:
Drug: Esomeprazole 40mg — Use in a drug combination for H. pylori eradication
Drug: Clarithromycin 500mg — Use in a drug combination for H. pylori eradication
Drug: Metronidazole 500 mg — Use in a drug combination for H. pylori eradication
  Arms: Empirical concomitant therapy
Drug: Amoxicillin 1000 MG — Use in a drug combination for H. pylori eradication
Drug: Levofloxacin 500mg — Use in a drug combination for H. pylori eradication
  Arms: Genotypic resistance-guided triple therapy
Drug: Rifabutin 150 MG — Use in a drug combination for H. pylori eradication
  Arms: Genotypic resistance-guided triple therapy

SUMMARY:
This study aims to investigate the efficacy of a 7-day genotypic resistance-guided triple therapy, compared with empirical concomitant therapy, for first-line eradication of H. pylori.

DETAILED DESCRIPTION:
Empiric eradication of H. pylori becomes steadily more challenging because of increasing antibiotic resistance. In high-resistance countries where bismuth and/or tetracycline are unavailable (eg; Greece), non-bismuth quadruple therapies are currently recommended as first-line therapeutic options; however, eradication rates >95% are infrequently achieved and even >90% are disputed. Antimicrobial susceptibility-guided therapy is a promising alternative in order to maintain high therapeutic efficacy. However, traditional culture-based susceptibility testing methods have several shortcomings, including they are time-consuming and they do not 100% reflect in vivo eradication. Recent guidelines also recommend the use of molecular testing for evaluation of H. pylori antibiotic susceptibility. Nevertheless, the efficacy of genotypic resistance-guided treatment of H. pylori has been seldom appraised. Therefore, the investigators conducted this prospective randomized controlled trial aiming to investigate the efficacy of a 7-day genotypic resistance-guided triple therapy, compared with empirical concomitant therapy, for first-line eradication of H. pylori.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive outpatients aged ≥18 years with documented H. pylori infection. Mental and legal ability to provide written informed consent.

Exclusion Criteria:

* previous history of H. pylori eradication therapy
* history of allergies to the medications used
* previous esophageal or gastric surgery
* serious systemic disease
* pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Rate of H. pylori eradication | At least 6 weeks after treatment completion
  Rate of H. pylori eradication by intention to treat/per protocol in each group at least 6 weeks after treatment completion using the urea breath test.

SECONDARY OUTCOMES:
Rate of adverse effects | At least 6 weeks after treatment completion
  Adverse events were investigated by means of a structured clinical interview immediately after the completion of therapy. The subjects were asked to grade the severity of adverse events according to their influence on daily activities, experienced as "mild" (transient and well tolerated), "moderate" (causing discomfort and partially interfering with daily activities), or "severe" (causing considerable interference with daily activities).
Compliance rates | At least 6 weeks after treatment completion
  Drug compliance was determined by counting unused medication. For this purpose, any tablet that was not consumed was brought back to the clinic for pill count. Poor compliance was defined as taking less than 80% of the total medication prescribed.

CONTACTS AND LOCATIONS:
Locations (1):
- Konstantopoulio-Patision General Hospital, Athens, Nea Ionia, Greece

IPD SHARING:
Plan to Share IPD: No